CLINICAL TRIAL: NCT04525144
Title: Evaluating the Role of EGb 761 in the Syndrome of Mild Cognitive Impairment With Concomitant Cerebrovascular Disease (MCI + CVD)
Brief Title: EGb 761 in the Syndrome of MCI With Concomitant CVD
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Neuroscience Institute (Other)
Collaborators: Dr. Willmar Schwabe GmbH & Co. KG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EGB-MCI
Record Dates: First submitted 2020-08-20; First posted 2020-08-25 (Actual); Last update posted 2022-11-17 (Actual); Status verified 2022-11

CONDITIONS: Mild Cognitive Impairment; Cerebrovascular Disease
MeSH Terms: conditions — Cognitive Dysfunction; Cerebrovascular Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tebonin Forte (Experimental): Treatment: 120mg, twice a day, 52 weeks
  Interventions: Drug: Tebonin Forte
- Control (No Intervention): No Treatment

INTERVENTIONS:
Drug: Tebonin Forte — Dietary supplement: Gingko biloba EGb 761
  Arms: Tebonin Forte

SUMMARY:
EGb 761 has been demonstrated to be useful in improving cognitive and global clinical outcomes in patients with cognitive impairment or dementia, when administered at a daily dosage of 240mg in randomised controlled trials through several neuroprotective mechanisms of action. The study aims to determine the efficacy and safety profile of EGb 761 as a prescribed clinical drug for patients with MCI + CVD.

DETAILED DESCRIPTION:
EGb 761 has been demonstrated to be useful in improving cognitive and global clinical outcomes in patients with cognitive impairment or dementia, when administered at a daily dosage of 240 mg in randomised controlled trials through several neuroprotective mechanisms of action.

The study aims to determine the efficacy and safety profile of EGb 761 as a prescribed clinical drug for patients with MCI + CVD. This study is an open label 52-weeks study in subjects who have both MCI (based on the Petersen criteria and Albert MS criteria) and CVD. Eligibility for enrolment will be assessed initially at a screening visit, which is to occur within 42 days of baseline. 134 male and female subjects will participate and 67 of the 134 will receive the drug.

Subjects will be randomized to the EGB 761 arm and control arm in a 1:1 ratio using a block randomization method in groups of 4 subjects using an automated randomization software. The study will allow generating data in an Asian and multi-racial population and allows physicians to offer clinically efficacious and alternative treatment for patients with MCI + CVD.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have been diagnosed with MCI based on the Petersen criteria and Albert MS criteria
* Patients who have a Global Clinical Dementia Rating Score of 0.5
* Patients aged 45 to 85 years at study entry
* Patients who are literate and able to complete the cognitive evaluations in the opinion of the investigators
* Patients with the presence of CVD, defined as the presence of white matter hyperintensities (WMH) of Fazekas grade 2 or 3 on MRI brain imaging (done up to 12 months prior to recruitment) or CT scans for patients contraindicated from MRI scans
* Patients who provide written informed consent to participate in the study

Exclusion Criteria:

* Participants should not be receiving antidepressants, antipsychotics, benzodiazepines, acetylcholinesterase inhibitors or NMDA antagonists during the study. Additionally, contraindications for EGb 761 as given in the local prescribing information/Summary of Product Characteristics (SmPC) should be observed.

Ages: 45 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Estimated)
Dates: Start 2020-10-26 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Alzheimer's Disease Assessment Scale-Cognitive 13 (ADAS-Cog 13) | 52 weeks
  Cognitive assessment
Clinical Dementia Rating Sum of Boxes Scores (CDR-SOB) | 52 weeks
  Functional assessment

SECONDARY OUTCOMES:
Visual Cognitive Assessment Tool (VCAT) | 52 weeks
  Cognitive assessment
Mild Behavioural Impairment Checklist (MBI-C) | 52 weeks
  Behavioral assessment

CONTACTS AND LOCATIONS:
Overall Officials: Kok Pin Ng, Principal Investigator — National Neuroscience Institute
Locations (1):
- National Neuroscience Institute, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Herrschaft H, Nacu A, Likhachev S, Sholomov I, Hoerr R, Schlaefke S. Ginkgo biloba extract EGb 761(R) in dementia with neuropsychiatric features: a randomised, placebo-controlled trial to confirm the efficacy and safety of a daily dose of 240 mg. J Psychiatr Res. 2012 Jun;46(6):716-23. doi: 10.1016/j.jpsychires.2012.03.003. Epub 2012 Mar 27. PMID 22459264
- [Background] Muller WE, Eckert A, Eckert GP, Fink H, Friedland K, Gauthier S, Hoerr R, Ihl R, Kasper S, Moller HJ. Therapeutic efficacy of the Ginkgo special extract EGb761(R) within the framework of the mitochondrial cascade hypothesis of Alzheimer's disease. World J Biol Psychiatry. 2019 Mar;20(3):173-189. doi: 10.1080/15622975.2017.1308552. Epub 2017 May 2. PMID 28460580
- [Background] Gavrilova SI, Preuss UW, Wong JW, Hoerr R, Kaschel R, Bachinskaya N; GIMCIPlus Study Group. Efficacy and safety of Ginkgo biloba extract EGb 761 in mild cognitive impairment with neuropsychiatric symptoms: a randomized, placebo-controlled, double-blind, multi-center trial. Int J Geriatr Psychiatry. 2014 Oct;29(10):1087-95. doi: 10.1002/gps.4103. Epub 2014 Mar 16. PMID 24633934
- [Background] Ihl R, Bachinskaya N, Korczyn AD, Vakhapova V, Tribanek M, Hoerr R, Napryeyenko O; GOTADAY Study Group. Efficacy and safety of a once-daily formulation of Ginkgo biloba extract EGb 761 in dementia with neuropsychiatric features: a randomized controlled trial. Int J Geriatr Psychiatry. 2011 Nov;26(11):1186-94. doi: 10.1002/gps.2662. Epub 2010 Dec 7. PMID 21140383
- [Background] Yuan Q, Wang CW, Shi J, Lin ZX. Effects of Ginkgo biloba on dementia: An overview of systematic reviews. J Ethnopharmacol. 2017 Jan 4;195:1-9. doi: 10.1016/j.jep.2016.12.005. Epub 2016 Dec 7. PMID 27940086